CLINICAL TRIAL: NCT04192981
Title: A Phase I Study With Expansion Cohort of Concurrent GDC-0084 With Radiation Therapy for Patients With Solid Tumor Brain Metastases or Leptomeningeal Metastases Harboring PI3K Pathway Mutations
Brief Title: GDC-0084 With Radiation Therapy for People With PIK3CA-Mutated Solid Tumor Brain Metastases or Leptomeningeal Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Kazia Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-359
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases; Leptomeningeal Metastasis
Keywords: GDC-0084; Radiation; PIK3CA Mutations; 19-359
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis | interventions — GDC-0084

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Concurrent GDC-0084 with Radiation (Experimental): GDC-0084 in 3 + 3 dose-escalation in 3 cohorts: 45, 60, 75 mg daily, with a potential de-escalation cohort to 30mg, to determine MTD in combination with whole brain radiation therapy radiation therapy to 30Gy in 10 fractions. Once MTD is determined, 12 additional patients will be treated with GDC-0084 at MTD in combination with whole brain radiation therapy.
  Interventions: Drug: GDC-0084; Radiation: whole brain radiation therapy radiation

INTERVENTIONS:
Drug: GDC-0084 — GDC-0084 in 3 + 3 dose-escalation in 3 cohorts: 45, 60, 75 mg daily
Radiation: whole brain radiation therapy radiation — 30Gy in 10 fractions

SUMMARY:
This study will test the safety of the study drug, GDC-0084, in combination with radiation therapy in people who have solid tumor brain metastases or leptomeningeal metastases. All participants will have cancer with a PIK3CA mutation. The researchers will test increasing doses of GDC-0084 to find the highest dose that causes few or mild side effects in participants. The study will also try to find out if the combination of the study drug with radiation is effective against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor malignancies harboring PIK3CA mutations which include mutations in any of the following genes: PIK3CA, PIK3CB, PIK3CD, PIK3CG, PIK3R1, PIK3R2, PIK3R3, PIK3C2G, PIK3C3, INPP4A, INPP4B, INPPL1, INPP5D, PTEN, AKT1, AKT2, AKT3, and MTOR.
* Brain metastases and/or leptomeningeal metastases involving the brain demonstrated by MR imaging of the brain. For patients with brain metastases, measurable lesion by RANO-BM is required28. Patients with spine leptomeningeal metastases are eligible for the study if they have leptomeningeal metastases of the brain demonstrated by MRI imaging of the brain.
* KPS ≥ 70
* Age ≥ 18 years
* Able to provide informed consent.
* If a patient is on corticosteroid, he/she must be on a stable daily dose of < 4mg dexamethasone or equivalent. Patient does not need to be given corticosteroid as prophylaxis if not clinically indicated.
* No limit to prior therapies with the last systemic therapy ≥ 1 week from initiation of protocol therapy. Systemic therapy can resume after completion of protocol DLT assessment period.
* Patients with prior SRS are eligible, provided that there are new, non-irradiated brain lesions or leptomeningeal metastases. Patients must be ≥ 3 months post prior cranial radiation therapy.
* Patients with seizure history related to brain metastases or leptomeningeal metastases controlled on antiepileptic medications are eligible.
* Patient at reproductive potential must agree to practice an effective contraceptive method
* Patient must be able to swallow and retain oral medication
* Adequate organ function as assessed by laboratory tests.
* Adequate bone marrow function

  * Hemoglobin ≥ 8g/dL
  * Absolute neutrophil count ≥1,000/mm^3
  * Platelet count ≥ 100,000/mm^3
* Adequate liver function

  * Bilirubin ≤1.5 times upper limit normal (ULN)
  * AST and ALT ≤ 2.5 times ULN
  * Alkaline phosphatase ≤ 2 times ULN
* Adequate renal function ° BUN and Creatinine ≤ 1.5 times ULN

Exclusion Criteria:

* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects tissue tolerances
* Patients with brain metastases eligible for single fraction stereotactic radiation therapy
* Serious medical co-morbidities precluding radiotherapy
* Insulin-treated diabetes; subjects with diabetes or impaired glucose tolerance that is not treated with insulin may be enrolled
* QT interval ≥ 450 msec on EKG
* Cardiac dysfunction defined as: myocardial infarction within 6 months of study entry, NYHA Class II/III/IV heart failure, unstable angina or unstable cardiac arrhythmias
* Known hypersensitivity or intolerance to GDC-0084 or to any other inhibitor of the PI3K/ Akt/ mTOR pathway
* Past medical history of interstitial lung disease, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease
* Subject receiving any medications or substances that are moderate and/or potent enzyme inducers or inhibitors which may have an effect on the metabolism of GDC-0084.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 1 year
  Four dose levels will be examined and the maximum tolerated dose (MTD) will be identified.
  The standard 3+3 dose-escalation scheme for this study is as follows. Patients will be accrued to the study in cohorts of 3. For any given dose an initial cohort of 3 patients will be treated at that dose.The dose level will be escalated if none of the 3 exhibits any dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
local recurrence rate | 1 year
  For patients with brain metastases, response determination will be determined using Response Assessment in Neuro-Oncology Brain Metastases criteria28. For patients with leptomeningeal metastases, response assessment will be determined by investigator based on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Imber, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - BAPTIST ALLIANCE - MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York
  - University of Washington (Data Collection AND Data Analysis), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm